CLINICAL TRIAL: NCT01502124
Title: Norditropin® and Norditropin® Cartridges: An Open-Label, Randomized, Comparative Safety and Efficacy Trial in Children With Growth Hormone Deficiency
Brief Title: Safety and Efficacy of Somatropin in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGH-2124
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lyophilized (Active Comparator)
  Interventions: Drug: somatropin
- Liquid (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Injected subcutaneously 7 times per week after reconstitution with liquid buffer prior to use. Dose level of 0.024-0.050 mg/kg at the discretion of the practicing paediatric endocrinologists
  Arms: Lyophilized
Drug: somatropin — Injected subcutaneously 7 times per week. Dose level of 0.024-0.050 mg/kg at the discretion of the practicing paediatric endocrinologists
  Arms: Liquid

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to evaluate the safety profiles of Norditropin® (lyophilized somatropin) and Norditropin® cartridges (liquid somatropin) in children with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of short stature (height maximum 2 standard deviations of mean for age and gender) or inadequate growth deemed secondary to growth hormone deficiency (GHD)
* Naïve to growth hormone therapy

Exclusion Criteria:

* Known or suspected allergy to the trial product or related products
* Growth retardation attributable to causes other than GHD. Growth retardation attributable to diabetes mellitus, inborn errors of metabolism, primary bone disease, chromosomal disorders or disease of the genitourinary, cardiopulmonary, gastrointestinal or central nervous system; bone marrow transplantation or any syndrome known to give short stature (examples are: Prader-Willi Syndrome, Russell-Silver Syndrome, Turner Syndrome, Noonan Syndrome)
* Intrauterine growth retardation: birth weight below 3rd percentile, adjusted for gestational age
* Pregnancy or the intention to become pregnant
* Breast-feeding
* Administration of other growth-altering medication

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2001-05-08 (Actual); Primary Completion 2003-03-05 (Actual); Study Completion 2003-03-05 (Actual)

PRIMARY OUTCOMES:
Adverse events (especially injection site reactions)
Serious adverse events

SECONDARY OUTCOMES:
IGF-1 (Insulin-like growth factor 1) concentration
IGFBP-3 (Insulin-like growth factor binding protein 3) concentration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (18):
- United States (18):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Wilmington, Delaware
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Manhasset, New York
  - Novo Nordisk Investigational Site, Akron, Ohio
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Seattle, Washington

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com